CLINICAL TRIAL: NCT02697422
Title: Vet COACH (Veteran Peer Coaches Optimizing and Advancing Cardiac Health)
Brief Title: Veteran Peer Coaches Optimizing and Advancing Cardiac Health
Acronym: Vet-COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 14-063
Record Dates: First submitted 2016-02-16; First posted 2016-03-03 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Disease (CVD); Hypertension; Hyperlipemia; Obesity
Keywords: Smoking (tobacco use); Peer health coach; Systolic blood pressure; Framingham Cardiovascular risk score; Lipid; Health related quality of life; Health care utilization; Medication adherence; Physical activity; Nutrition; Alcohol use; Stress management
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Hyperlipidemias; Obesity; Smoking; Tobacco Use; Patient Acceptance of Health Care; Medication Adherence; Motor Activity; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of two groups--the control or intervention group- in parallel for the duration of the study.
Masking Description: N/A; No masking will occur in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer health coach intervention group (Experimental): Eligible participants will be randomly assigned to receive a home-visit peer health coach intervention to promote health outcomes and behavior change among Veterans with multiple cardiovascular disease (CVD) risk factors.
  Interventions: Other: Community-based peer health coach intervention
- Control group (No Intervention): Participants who meet the same eligibility criteria as participants in the intervention group will be randomly assigned to receive no intervention. Participants will continue to receive their regular, usual primary care.

INTERVENTIONS:
Other: Community-based peer health coach intervention — The focus of the peer health coach intervention will be to deliver brief health messages, discuss goal setting, and action planning around health behavior changes shown to decrease CVD risk (for instance, healthy diet, regular to moderate-intensity physical activity, and quitting smoking).
  Other Names: Vet-Coach intervention
  Arms: Peer health coach intervention group

SUMMARY:
The purpose of this study is to test if having a Veteran peer health coach will improve blood pressure control among Veterans with high blood pressure and at least one other Cardiovascular disease (CVD) risk factor. The intervention will deliver brief health messages, discuss goal setting, and action planning around health behavior changes shown to decrease CVD risk, including healthy diet, regular to moderate-intensity physical activity, and smoking cessation. Facilitators, barriers, and costs of the intervention will be determined.

DETAILED DESCRIPTION:
The Vet-COACH study is a peer health coaching program to help reduce Cardiovascular disease (CVD) risk among Veterans. The goal of the study is to test the effectiveness of a home-visit peer health coach intervention to promote health outcomes and behavior change among Veterans with multiple CVD risk factors with a hybrid type 1 implementation study. The study will focus on Veterans with poorly controlled hypertension and at least one other CVD risk factor to target a high risk population.

The study will conduct a randomized controlled trial to enroll n=400 Veterans to compare a peer health coach intervention consisting of home visits, telephone support, and linkages to appropriate community-based and clinic resources compared to usual VHA primary care. The primary outcome is reduction in systolic blood pressure from baseline to follow-up at 1-year. Secondary outcomes include a reduction in Framingham Cardiovascular risk score, individual cardiovascular risks (tobacco use, lipids), health related quality of life, and health care use. The investigators will also assess the effects of the peer health coach intervention on intermediate outcomes including social support, patient activation, patient/provider communication and health behaviors (e.g. medication adherence, physical activity, nutrition, alcohol use, and stress management). The cost of the intervention will be assessed to inform feasibility for future studies, determine Veteran and staff satisfaction with the intervention, and identify barriers and facilitators to adoption.

Note, the intermediate outcomes were not prespecified in the protocol for evaluation and were not specified in the grant, protocol paper, or in our SAP as outcomes and were removed from results analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Veteran
* Have > 1 visit to VA Puget Sound Health Care Center(Seattle or American Lake VA) primary care or women's clinic in the past year
* Poorly controlled hypertension (> 150/90 mmHg)
* At least one other CVD risk (including overweight or obesity, body mass index > 25 kg/m2, tobacco use, hyperlipidemia LDL-c > 130 mg/dL)

Exclusion Criteria:

* Hospitalization in the past 3 months for cardiovascular-related conditions (IHD, Cerebral Vascular Accident [CVA], PVD)
* Severe illness that precludes lifestyle program, end-stage renal disease (ESRD) on dialysis
* Nursing home resident, homeless
* Severe cognitive impairment
* Receiving home-based primary care (including VA Home Tele-Health and patients who received palliative care or are enrolled in hospice care)

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin M. Nelson, MD MSHS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will adhere to all VA 1200.12 policies to protect individual privacy & confidentiality of data. Data will be made available outside VA in response to a properly prepared Freedom of Information Act request submitted & evaluated by the VA Puget Sound FOIA Officer, or as passed down to the facility.
  A unique study ID will label all data records to allow validation of results, but prevent data from being linked to individuals. Records across data sets can be cross-referenced using the study ID to verify accuracy of publication results. Research publications will be made available to the public via the National Library of Medicine PubMed Central website within one year after publication date(s). A Limited Dataset will be created & shared pursuant a Data Use Agreement that appropriately limits use of the dataset & prohibits recipients from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.

REFERENCES:
- [Result] Nelson K, Fennell T, Gray KE, Williams JL, Lutton MC, Silverman J, Jain K, Augustine MR, Kopf W, Taylor L, Sayre G, Vanderwarker C. Veteran peer Coaches Optimizing and Advancing Cardiac Health (Vet-COACH); design and rationale for a randomized controlled trial of peer support among Veterans with poorly controlled hypertension and other CVD risks. Contemp Clin Trials. 2018 Oct;73:61-67. doi: 10.1016/j.cct.2018.08.011. Epub 2018 Aug 29. PMID 30172037
- [Result] Nelson KM, Taylor L, Williams JL, Rao M, Gray KE, Kramer CB, Epler E, Fennell T. Effect of a Peer Health Coaching Intervention on Clinical Outcomes Among US Veterans With Cardiovascular Risks: The Vet-COACH Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2317046. doi: 10.1001/jamanetworkopen.2023.17046. PMID 37278999
- [Derived] Kramer CB, Nelson KM, Sayre G, Williams JL, Spruill L, Fennell T, Gray KE, Weiner BJ, Fan V, Jones-Smith J, Rao M. "Veteran to Veteran, There's Automatically a Trust": A Qualitative Study of Veterans' Experiences in a Peer Health-Coaching Program for Hypertension. AJPM Focus. 2024 Jul 3;3(6):100257. doi: 10.1016/j.focus.2024.100257. eCollection 2024 Dec. PMID 39415799
- See also: published standardized scoring system for the SF-12 — https://www.researchgate.net/publication/242636950_SF-12_How_to_Score_the_SF-12_Physical_and_Mental_Health_Summary_Scales

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer Health Coach Intervention Group | Control Group
Started | 134 | 130
Completed | 108 | 117
Not Completed | 26 | 13
Not completed — Declined exit survey | 9 | 2
Not completed — Lost to Follow-up | 13 | 8
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Exit survey data lost | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Health Coach Intervention Group | Control Group | Total
Number analyzed (Participants) | 134 | 130 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.7) | 60.9 (9.8) | 60.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 35
  Male | 113 | 116 | 229
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 67 | 56 | 123
  Black, non-Hispanic | 37 | 36 | 73
  Multiracial | 13 | 17 | 30
  Hispanic | 7 | 10 | 17
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 137.1 (16.4) | 135.1 (19.6) | 136 (18.0)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 80.9 (9.6) | 81.3 (11.3) | 81.1 (10.48)
Hypertension Stage [Count of Participants; unit: Participants]
  Normal (<120/80 mmHg) | 13 | 28 | 41
  Elevated (>=120/80 mmHg) | 24 | 16 | 40
  Stage 1 (>=130/90 mmHg) | 65 | 52 | 117
  Stage 2 (>=140/90 mmHg) | 32 | 34 | 66
Framingham risk score [Mean (Standard Deviation); unit: percentage of CVD risk] — FRS score is determined according to FRS algorithms, which include age, total and high-density lipoprotein cholesterol, systolic blood pressure, treatment for hypertension, diabetes, and cigarette smoking. Risk is considered low if the FRS is less than 10% (indicating a better outcome), moderate if it is between 10% -19%, and high if it is 20% or higher indicating a worse outcome.
  percentage of CVD risk | .22 (.16) | .26 (.17) | .24 (.17)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (5.8) | 31.9 (6.3) | 31.8 (6.1)
CVD Risk: BMI category [Count of Participants; unit: Participants]
  Overweight (BMI>= 25 kg/m2) | 125 | 119 | 244
  Obese (BMI>= 30 kg/m2) | 73 | 76 | 149
CVD Risk: Current Smoker Status [Count of Participants; unit: Participants] | 21 | 29 | 50
CVD Risk: Low density lipoprotein (LDL-c) cholesterol [Mean (Standard Deviation); unit: mg/dL] | 107.0 (38.6) | 112.4 (38.7) | 109.6 (38.7)
Health-related quality of life (HRQoL) mental health mental health component summary (MCS) [Mean (Standard Deviation); unit: units on a scale] — Health-related quality of life is measured by the Medical Outcomes Study 12-item measure (SF-12). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
  units on a scale | 46.9 (11.7) | 47.4 (11.9) | 47.1 (11.8)
Health-related quality of life (HRQoL) physical health component summary (PCS) [Mean (Standard Deviation); unit: units on a scale] — Health-related quality of life is measured by the Medical Outcomes Study 12-item measure (SF-12). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
  units on a scale | 39.6 (10.6) | 38.9 (10.6) | 39.3 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change in systolic blood pressure (SBP) from baseline to 12-months. Blood pressure readings were obtained using standard procedures with a blood pressure monitor to obtain a mean SBP score of 3 blood pressure measurements. An increased reduction in mean SBP indicates a better outcome.
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
mm Hg | -3.32 [-6.88 to 0.23] | -0.40 [-4.20 to 3.39]
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

2. Secondary Outcome: Framingham Cardiovascular Risk Score (FRS)
Description: Framingham Cardiovascular risk score (FRS) indicates/measures mean risk of a cardiovascular event in the next 10 years (CVD risk). A subscale range of a minimum score of 0% and maximum score of 30% were used to measure a reduction in FRS scores. FRS algorithms include age, total and high-density lipoprotein cholesterol, systolic blood pressure, treatment for hypertension, diabetes, and cigarette smoking. (Risk is considered low if the FRS is less than 10% (indicating a better outcome), moderate if it is between 10% -19%, and high if it is 20% or higher indicating a worse outcome).
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (95% Confidence Interval); unit: percentage of CVD risk
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
percentage of CVD risk | -0.01 [-0.03 to 0.004] | -0.01 [-0.03 to 0.004]
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

3. Secondary Outcome: Body Mass Index (BMI)
Description: Body Mass Index (BMI) are measured as an individual cardiovascular risk. Measurements will be initially recorded in height (feet/inches), and weight (pounds/ ounces, which will be converted to weight in kilograms and height in meters. BMI is calculated as kg/m^2.
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
kg/m^2 | -0.04 [-0.48 to 0.40] | 0.10 [-0.3 to 0.5]
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

4. Secondary Outcome: Current Tobacco Use
Description: Current tobacco use was reported as a binary (YES/NO) outcome based on responses from the Behavioral Risk Factor Surveillance System (BRFSS) measured tobacco use. Current cigarette smoking status and tobacco use ("chewing tobacco, snuff or snus") and frequency of use were measured on a three point scale: "Every day" (worse outcome); "Some days", and "Not at all" (better outcome). Current tobacco use included individuals who reported having smoked at least 100 cigarettes in their entire life (Yes or No) and reported smoking cigarettes now ("Every day" or "Some days"). Differences in primary and secondary outcomes between intervention and control groups were calculated using logistic regression.
Time Frame: Current tobacco use measured at Baseline and Follow up at one year
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
Participants | 21 | 29
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Smoker/tobacco use results were calculated using logistic regression. A P value of .90 was found comparing smoking/tobacco use in intervention vs control participants. A difference was not reported between intervention and control because smoking/ tobacco use was a binary variable; Test type: Superiority; p = 0.90, Regression, Logistic — Smoker/tobacco use results were calculated using logistic regression

5. Secondary Outcome: Low Density Lipoprotein Cholesterol (LDL-c).
Description: Low density lipoprotein cholesterol (LDL-c) is measured as mg/dL. Lipoprotein cholesterol will be assessed as an individual cardiovascular risk and is based laboratory data of blood tests from VA CPRS medical records (when taken within 6 months of baseline and/or 1 year follow up appointment). If no lab data exits within this timeframe, blood was drawn.
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
mg/dL | -3.12 [-8.36 to 2.12] | -4.24 [-9.75 to 1.27]
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

6. Secondary Outcome: Change in Health-Related Quality of Life (HRQoL), Mental Component Summary Score
Description: 12-Item Short Form Health Survey (SF-12) Mental Component Summary: Summary scores for vitality, mental health, social functioning, and role-emotional. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning Scaling scores are assessed using published standardized scoring system procedures for the SF-12.
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
points | 2.19 [0.26 to 4.12] | -1.01 [-2.91 to 0.88]
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

7. Secondary Outcome: Change in Health-Related Quality of Life (HRQoL), Physical Component Summary Score (PCS)
Description: 12-Item Short Form Health Survey (SF-12) Physical Component Summary: Summary scores for general health, physical functioning, role-physical, and bodily pain. Scores range from a minimum score of 0 to a maximum score of 100, with higher scores indicating better physical and mental health functioning Scaling scores are assessed using published standardized scoring system for the SF-12.
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (95% Confidence Interval); unit: points on a 0-100 scale
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
points on a 0-100 scale | 1.02 [-0.73 to 2.77] | 0.72 [-0.82 to 2.27]
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

8. Secondary Outcome: Number of Hospitalizations
Description: Health care hospitalization utilization are measured using VA administrative data.
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
visits | 0.16 (0.53) | 0.13 (0.47)
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

9. Secondary Outcome: Number of Emergency Room (ER) Visits
Description: Health care emergency room (ER) utilization are measured using VA administrative data.
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
visits | 0.86 (1.37) | 0.86 (1.66)
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

10. Secondary Outcome: Number of Outpatient Clinic/Primary Care Visits
Description: Outpatient clinic/primary care utilization are measured using VA administrative data.
Time Frame: Baseline to follow-up at 1 year
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Peer Health Coach Intervention Group | Control Group
Number analyzed (Participants) | 134 | 130
visits | 0.40 (0.89) | 0.55 (1.35)
Statistical Analysis 1: Comparison: Peer Health Coach Intervention Group vs Control Group; Test type: Superiority; p = 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: Baseline to follow up at 1 year
Description: Study intervention posed minimal risk to all participants. Deaths were assessed and determined to be unrelated to the study intervention.
Arm/Group | Peer Health Coach Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/134 | 1/130
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/130
Other Adverse Events (participants affected / at risk) | 0/134 | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT02697422/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT02697422/SAP_001.pdf